CLINICAL TRIAL: NCT00531492
Title: Randomized Controlled Trial of Continuous Skin to Skin Care (Technique Kangourou: TK) for Low Birth Weight (LBW) Infants and Their Mothers at University Hospital Center of Mahajanga (Centre Hospitalier Universitaire de Mahajanga: CHUM), Madagascar
Brief Title: Efficacy of Continuous Skin to Skin Care (Technique Kangaroo: TK) After Birth for Low Birth Weight (LBW) Infants and Their Mothers in Developing Countries
Acronym: EtudeTK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Advanced Studies on International Development (Other)
Collaborators: St.Luke's Life Science Institute, Tokyo, Japan (Unknown)
Responsible Party: Principal Investigator, Shuko Nagai, Groupe d'Etude de la Technique Kangourouà, Foundation for Advanced Studies on International Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FASID-06-CE-56
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Low Birth Weight
Keywords: Maternal and child health; Developing country; Skin to skin care; Newly born low birth weight infants and their mothers; (Delivery at University Hospital Center, Mahajanga, Madagascar)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Behavioral: TK as soon as possible within 24 hours after birth
- B (Active Comparator)
  Interventions: Other: Conventional care

INTERVENTIONS:
Behavioral: TK as soon as possible within 24 hours after birth — Start TK as soon as possible within 24 hours after birth
  Arms: A
Other: Conventional care — Start conventional care (At first use incubator, and start TK when the infants and mother are completely settled and ready)
  Arms: B

SUMMARY:
The purpose of this study is to examine the efficacy of Technique Kangourou (TK) between low birth weight (LBW) infants and their mothers started as soon as possible within 24 hours after birth in developing country.

For the purpose of this study, TK is defined as skin-to-skin direct and continuous (24 hours) contact between LBW infants and their mothers or any other people who substitute mothers.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight (BW) < 2500g
* Delivery at maternity of CHUM (Birth < 24 hours)
* Without serious congenital malformation
* Sat O2 >=95％, HR > 100 / min, RR < 60 / min, Capillary refilling time < 3 sec
* The mother and the family are motivated to practice TK.
* The mother and the family available to practise TK should be healthy.

Exclusion Criteria:

* Apnea of prematurity >20 sec
* With intravenous infusion

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Mortality within 28 days after birth | within 28 days after birth

SECONDARY OUTCOMES:
Mobility within 28 days after birth | within 28 days after birth
Mortality and Mobility within 28 days after birth | within 28 days after birth
Difference of (Baby's) loss in weight within 2 days | within 2 days
Difference of (Baby's) Body weight of 14th day after birth | 14th day after birth
Difference of (Baby's) Body weight of 28th day after birth | 28th day after birth
Incidence of hypothermia during hospitalisation and (or) during outpatient department （lower than 35.5℃） | Within 28 days after birth
Incidence of bradycardia or tachycardia during hospitalisation (HR <100, or>180 /min) | within 28 days after birth
Incidence of apnea during hospitalisation (> 20 sec) | within 28 days after birth
Incidence of desaturation during hospitalisation ( <87%) | within 28 days after birth
Length of hospitalisation | within 28 days after birth
Discharge within 7days after birth | within 7days after birth
Mobility within 6 months or 1 year after birth | within 6 months or 1 year
Mortality and Morbility within 6 months or 1 year after birth | within 6 months or 1 year
Mortality within 6 months or 1 year after birth | within 6 months or 1 year
Incidence of hyperthermia during hospitalisation and (or) outpatient department （upper than 37.5℃） | Within 28 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Shuko Nagai, MD, Principal Investigator — Groupe d'Etude de la Technique Kangourouà Mahajanga, Madagascar
Locations (1):
- University Hospital Center of Mahajanga (Centre Hospitalier Universitaire de Mahajanga: CHUM),, Mahajanga, Mahajanga, Madagascar

REFERENCES:
- [Result] Nagai S, Andrianarimanana D, Rabesandratana N, Yonemoto N, Nakayama T, Mori R. Earlier versus later continuous Kangaroo Mother Care (KMC) for stable low-birth-weight infants: a randomized controlled trial. Acta Paediatr. 2010 Jun;99(6):827-35. doi: 10.1111/j.1651-2227.2009.01676.x. Epub 2010 Jan 27. PMID 20121708
- [Result] Nagai S, Yonemoto N, Rabesandratana N, Andrianarimanana D, Nakayama T, Mori R. Long-term effects of earlier initiated continuous Kangaroo Mother Care (KMC) for low-birth-weight (LBW) infants in Madagascar. Acta Paediatr. 2011 Dec;100(12):e241-7. doi: 10.1111/j.1651-2227.2011.02372.x. Epub 2011 Jun 23. PMID 21635363